CLINICAL TRIAL: NCT02214498
Title: Treatment of HYpertension: Morning Versus Evening
Acronym: THYME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Jorie Versmissen, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014_THYME
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Essential Hypertension
Keywords: Dipper; Non-dipper; Chronopharmacology
MeSH Terms: conditions — Essential Hypertension | interventions — Vaseretic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enalapril/hydrochlorothiazide (Active Comparator): This arm will start with six weeks of administration of enalapril/hydrochlorothiazide in the evening and placebo in the morning, followed by six weeks of active treatment in the morning and placebo in the evening
  Interventions: Drug: Enalapril/hydrochlorothiazide; Drug: Placebo
- Placebo (Placebo Comparator): This arm will start with six weeks of morning administration of enalapril/hydrochlorothiazide in the morning and placebo in the evening, followed by six weeks of placebo in the morning and active treatment in the evening
  Interventions: Drug: Enalapril/hydrochlorothiazide; Drug: Placebo

INTERVENTIONS:
Drug: Enalapril/hydrochlorothiazide — The intervention implies that morning and evening administration of enalapril/hydrochlorothiazide will be compared
  Other Names: To be determined
Drug: Placebo

SUMMARY:
Rationale:

The nocturnal blood pressure mean is an independent and stronger predictor of cardiovascular disease (CVD) risk than either daytime office, awake or 24hour mean blood pressure. In general, when nocturnal blood pressure does not decline CVD risk is higher, usually referred to as "dippers" versus "non-dippers". Evening administration of treatment might lower nocturnal blood pressure more effectively than morning administration, which is most commonly advised.

The main hypothesis of this study is that evening administration of antihypertensive medication might resume the dipping pattern in non-dippers and as a consequence might reduce CVD risk more than morning administration.

Primary objective (in short):

-to prove that evening administration of enalapril/hydrochlorothiazide in non-dippers can resume a dipping blood pressure pattern in non-dippers

Study design: A double-blind placebo-controlled cross-over study Each person will use for one period of six weeks enalapril/hydrochlorothiazide in the morning and placebo in the evening, and one period of six weeks the other way around

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension
* Stable blood pressure on treatment with Angiotensin Converting Enzyme Inhibitor (ACEI) or Angiotensin II Receptor Blocker (ARB) and hydrochlorothiazide
* Age between 18 and 85 years
* WHO performance status 0-1
* Available for a time period of 15 weeks
* Written informed consent
* Dippers: Nocturnal blood pressure fall of 10-20% of daytime values.20
* Non-dippers: -Nocturnal blood pressure fall of <10% of daytime values

Exclusion Criteria:

* secondary cause of hypertension
* use of ARB because of intolerability (e.g. dry cough) of ACEI
* nocturnal blood pressure fall of >20% or rise
* renal insufficiency (GFR<60 ml/min)
* shift work
* pregnancy or wish to get pregnant
* use of other antihypertensive medication than ACEI, ARB, hydrochlorothiazide or a calcium channel blocker
* use of sleeping medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Average nocturnal blood pressure, percentage dipping and nadir of nocturnal blood pressure | 24 hours
  At the end of each treatment period of six weeks, a 24 hour ambulatory blood pressure measurement will be performed

SECONDARY OUTCOMES:
Percentage of nocturnal diastolic blood pressure measurements below 65 mm hg | 24 hours
  One safety issue on evening administration of antihypertensive treatment is that blood pressure might get too low. We will assess this especially in the dippers.
Urine: Sodium, potassium, protein, melatonin, creatinin | Two times within 24 hours at the end of six weeks of treatment according to one of the two regimes
  Excretion of sodium, potassium, protein and melatonin depend on the circadian clock. Therefore, differences between morning and evening administration of antihypertensive medication are tested
Plasma: enalapril, cortisol, melatonin, aldosterone, ACE activity, gene expression of clock genes | Moring of 24 hour blood pressure measurement after six weeks of treatment according to a certain regime

CONTACTS AND LOCATIONS:
Overall Officials: Jorie Versmissen, MD, PhD, Principal Investigator — Erasmus Medical Center; Teun Van Gelder, Prof, Study Director — Erasmus Medical Center; Eric Sijbrands, Prof, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands